CLINICAL TRIAL: NCT02792738
Title: Effect of Hypnosis on Dyspnea
Acronym: Hypnopnee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ADOREPS_3
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Healthy; Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hypnosis, visual distraction (Experimental): This is a crossover study in which each subject will be exposed to a 5 min phase of hypnotic suggestion and visual distraction.
  For hypnotic suggestion, subject will be invited to experience a pleasant memory . Indirect and permissive suggestion will be used.
  For visual distraction, subject will be watching the movie "la marche des empereurs"
  Interventions: Behavioral: hypnosis

INTERVENTIONS:
Behavioral: hypnosis

SUMMARY:
The purpose of this protocol is to test the effect of hypnosis on laboratory dyspnea.

DETAILED DESCRIPTION:
This is a study of permissive suggestion in two laboratory models of dyspnea ("work/effort", "air hunger"). Breathing discomfort rating induced by laboratory models of dyspnea will be assessed before, during and after hypnosis.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* pregnancy
* ongoing pain
* respiratory disease
* high levels of depression, panic disorder, or other significant mental health problems
* not fluent in french

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

PRIMARY OUTCOMES:
Subject rating of Breathing Discomfort (affective component of dyspnea) | continuous measurement for 5 minutes
  Subjects will rate breathing discomfort using a visual analog scale at baseline (pre-intervention), during the intervention (hypnosis/ visual distraction) and after intervention (recovery) while subject will be submitted to the laboratory model of dyspnea for 5 minutes (three runs of laboratory dyspnea (baseline, intervention and recovery).
Subject rating of dyspnea intensity (sensory component of dyspnea) | continuous measurement for 5 minutes
  Subjects will rate dyspnea intensity using a visual analog scale at baseline (pre-intervention), during the intervention (hypnosis/ visual distraction) and after intervention (recovery) while subject will be submitted to the laboratory model of dyspnea for 5 minutes (three runs of laboratory dyspnea (baseline, intervention and recovery).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie et Réanimation Médicale, Paris, France

IPD SHARING:
Plan to Share IPD: No